CLINICAL TRIAL: NCT05081960
Title: Evaluating the Vitamin K2 Status of Calcium-based Stone Formers
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Principal Investigator, Jennifer Bjazevic, Principal Investigator, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 119537
Record Dates: First submitted 2021-09-22; First posted 2021-10-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-08

CONDITIONS: Kidney Calculi; Calcium Oxalate Kidney Stones; Vitamin K 2; Human; Kidney Stone; Calcium Oxalate Urolithiasis; Calcium Phosphate Urolithiasis; Nephrolithiasis
Keywords: Kidney stone disease; Microbiota; Menaquinone; Vitamin K2; Matrix Gla protein; dp-ucMGP; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis, Calcium Oxalate; Nephrolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, fecal, and blood samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stone Formers: Individuals who have experienced at least one incidence of calcium-based kidney stones in the last 12 months
- Controls: Individuals who have never had a kidney stone in their lifetime.

SUMMARY:
This is an observation, single site-study with one study visit during which all data and samples will be collected. Study participants will be asked to provide blood, urine, and fecal samples so that the investigators may study the differences in the gut microbiota, vitamin K2 levels, and other parameters between participants who form kidney stones and those who do not.

DETAILED DESCRIPTION:
It is hypothesized that calcium-based stone formers will have an altered fecal gut microbiota compared to non-stone former controls. This altered microbiota will have a lower abundance of bacteria that produce menaquinones (vitamin K2), thus stone formers will also have a different blood menaquinone profile compared to controls. Ultimately, the different levels of menaquinones will result in increased inactive Matrix Gla protein (dp-ucMGP), which is a key protein that sequesters free calcium. To test this hypothesis, calcium-based stone former and non-stone forming controls will be recruited to a single site, observation study to collect urine, blood, and fecal samples. These samples will be used to determine dp-ucMGP levels, menaquinone profiles, the composition of the gut microbiota, and other parameters of interest.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, 18 - 65 years old
* No self-reported kidney stones during their lifetime (controls)
* Ultrasound examination confirming absence of kidney stones (controls)
* Have had at least 1 incidence of a clinically confirmed calcium-based kidney stone in the last 12 months (stone formers)
* Ability to collect a clean catch urine sample
* Prescription and over-the-counter drugs unchanged for ≥30 days
* Willingness to provide medical information, blood, urine, and fecal samples

Exclusion Criteria:

* Current, or within 30 days, use of antibiotics or antifungals
* Current, or within 30 days, use of vitamin K antagonists
* Current probiotic use or any use within 14 days of screening sample collection should be recorded
* A history or currently undergoing immunosuppressive drug therapy, chemotherapy, or radiation therapy 2021-06-29 1.0 Page 4 of 6
* Fecal incontinence
* History of disorder with abnormal calcium regulation such as hyperparathyroidism, active malignancy, or osteoporosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stone formers will be recruited from the Urology clinic or London and surrounding community. Controls will be recruited from the London and surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota composition of stone-formers and controls | At baseline only
  Fecal samples will be collected using out validated toilet paper method. Microbial DNA will be extracted and sequenced using next-generation sequencing.
Concentration of urine dp-ucMGP (dephosphorylated-uncarboxylated Matrix Gla Protein) | At baseline only
  dp-ucMGP will be quantified using an enzyme-linked immunosorbent assay
Concentration of blood dp-ucMGP (dephosphorylated-uncarboxylated Matrix Gla Protein) | At baseline only
  dp-ucMGP will be quantified using an enzyme-linked immunosorbent assay
Concentration of blood total osteocalcin (OC) | At baseline only
  Total OC will be quantified using an enzyme-linked immunosorbent assay
Concentration of blood undercarboxylated osteocalcin (ucOC) | At baseline only
  ucOC will be quantified using an enzyme-linked immunosorbent assay
Concentration of urine total osteocalcin (OC) | At baseline only
  Total OC will be quantified using an enzyme-linked immunosorbent assay
Concentration of urine undercarboxylated osteocalcin (ucOC) | At baseline only
  ucOC will be quantified using an enzyme-linked immunosorbent assay
Concentration of blood menaquinones (vitamin K2) - MK-4 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-7 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-8 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-9 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-10 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-11 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-12 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.
Concentration of blood menaquinones (vitamin K2) - MK-13 | At baseline only
  Menaquinones will be quantified using liquid chromatography with mass spectrometry or fluorescence.

SECONDARY OUTCOMES:
Concentration of blood fetuin A | At baseline only
  Fetuin A will be quantified using enzyme-linked immunosorbent assay
Concentration of urine fetuin A | At baseline only
  Fetuin A will be quantified using enzyme-linked immunosorbent assay
Percentage of blood Hemoglobin A1C (HbA1c) | At baseline only
  HbA1c will be quantified in the core laboratory as per established protocols
Total plasma calcium | At baseline only
  Calcium levels will be quantified in the core laboratory
Concentration of ionized calcium in blood | At baseline only
  Calcium levels will be quantified in the core laboratory
Concentration of blood albumin | At baseline only
  Albumin levels will be quantified in the core laboratory as per established protocols
Concentration of urinary γ-carboxyglutamic acid | At baseline only
  γ-carboxyglutamic acid will be quantified using high-performance liquid chromatography and normalized to creatinine
Concentration of urinary creatinine | At baseline only
  Creatinine will be quantified using high-performance liquid chromatography
Concentration of urinary oxalate | At baseline only
  Oxalate will be quantified using high-performance liquid chromatography and normalized to creatinine
Concentration of urinary phosphate | At baseline only
  Phosphate will be quantified in the core laboratory as per established protocols

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bjazevic, MD, Principal Investigator — Lawson Heath Research
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conly J, Stein K. Reduction of vitamin K2 concentrations in human liver associated with the use of broad spectrum antimicrobials. Clin Invest Med. 1994 Dec;17(6):531-9. PMID 7895417
- [Background] Fraser JD, Price PA. Lung, heart, and kidney express high levels of mRNA for the vitamin K-dependent matrix Gla protein. Implications for the possible functions of matrix Gla protein and for the tissue distribution of the gamma-carboxylase. J Biol Chem. 1988 Aug 15;263(23):11033-6. PMID 3042764
- [Background] Moe OW. Kidney stones: pathophysiology and medical management. Lancet. 2006 Jan 28;367(9507):333-44. doi: 10.1016/S0140-6736(06)68071-9. PMID 16443041
- [Background] Sato T, Schurgers LJ, Uenishi K. Comparison of menaquinone-4 and menaquinone-7 bioavailability in healthy women. Nutr J. 2012 Nov 12;11:93. doi: 10.1186/1475-2891-11-93. PMID 23140417
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Schurgers LJ, Vermeer C. Determination of phylloquinone and menaquinones in food. Effect of food matrix on circulating vitamin K concentrations. Haemostasis. 2000 Nov-Dec;30(6):298-307. doi: 10.1159/000054147. PMID 11356998
- [Background] Schurgers LJ, Vermeer C. Differential lipoprotein transport pathways of K-vitamins in healthy subjects. Biochim Biophys Acta. 2002 Feb 15;1570(1):27-32. doi: 10.1016/s0304-4165(02)00147-2. PMID 11960685
- [Background] Stanford J, Charlton K, Stefoska-Needham A, Ibrahim R, Lambert K. The gut microbiota profile of adults with kidney disease and kidney stones: a systematic review of the literature. BMC Nephrol. 2020 Jun 5;21(1):215. doi: 10.1186/s12882-020-01805-w. PMID 32503496
- [Background] Wei FF, Thijs L, Zhang ZY, Jacobs L, Yang WY, Salvi E, Citterio L, Cauwenberghs N, Kuznetsova T, E A Drummen N, Hara A, Manunta P, Li Y, Verhamme P, Allegaert K, Cusi D, Vermeer C, Staessen JA. The risk of nephrolithiasis is causally related to inactive matrix Gla protein, a marker of vitamin K status: a Mendelian randomization study in a Flemish population. Nephrol Dial Transplant. 2018 Mar 1;33(3):514-522. doi: 10.1093/ndt/gfx014. PMID 28340119
- [Background] Chmiel JA, Stuivenberg GA, Al KF, Akouris PP, Razvi H, Burton JP, Bjazevic J. Vitamins as regulators of calcium-containing kidney stones - new perspectives on the role of the gut microbiome. Nat Rev Urol. 2023 Oct;20(10):615-637. doi: 10.1038/s41585-023-00768-5. Epub 2023 May 9. PMID 37161031